CLINICAL TRIAL: NCT02629471
Title: Study of the Effects of Light Flashes on the Visual System
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Analyzing data
Sponsor: LightGuard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LG01
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2019-12

CONDITIONS: Light Flashing Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- response time due to light flashs pulses (Experimental): light flashing effects on response time to random target appearance
  Interventions: Behavioral: response time due to light flash pulses

INTERVENTIONS:
Behavioral: response time due to light flash pulses — light flash pulses effect on response time to random targets appearance

SUMMARY:
Background The goal of this study is to examine the human visual and cognitive performance under the effect of bright light pulses. Exposure to visual stimulation of such pulsation may interfere with cognitive function and at certain situations this may be noticeable and may interfere with our judgment and abilities. In some of them visual or cognitive impairment from exposure to bright light flashes may result in catastrophic outcome due to the high-risk situation e.g. road accidents. Ocular exposure to a bright light can result in profound momentary transitional loss of vision. The light sources employed for visual stimulation in this study will be restricted to the range consistent with "reversible effects" (e.g. glare and flash insensitivity or "flash blindness").

The impact of an exposure to bright light depends not only on the exposure level and frequency, but also on the exposed individual's activity, psychological state, adaptation level and visual task. Glare is primarily caused by the scattering of light within the eye due to the imperfect transparency of the optical components of the eye and to a lesser extent by diffuse light passing through the scleral wall or the iris. The scattered light overlays the retinal image, thus reducing visual contrast. Excessive glare may impair visual function and lead to temporary disability.

The above mentioned effects of exposure to light and pulsating light stimulus on the visual system and cognition were studied in detail by a number of groups. These studies indicate that the visual and cognition effects of pulsating light are a function of the following parameters: pulse duration, light intensity and pulse frequency.

DETAILED DESCRIPTION:
Study Purpose and Rationale The purpose of this study is to evaluate the cognitive effects of exposure to flashing light stimuli by measuring the response time and level of performance of healthy human subjects during exposure to light pulsations.

Study Design and methods:

1. Overall study design An open prospective study comprising of cognitive tests performed during and following exposure to bright flashing light stimuli.

   Pre and post -cognitive test (within 1 month after the test) ophthalmological tests will be conducted.
2. Study Participants A total of 60 subjects will be recruited for this study over a span of 3 months.

The subjects will volunteer to participate in the study. Flash Tests The subject will be positioned at a selected distance from a flashing unit and a screen on which different scenarios will be projected.

The subject will be exposed to the flashing light generated by the study device with various parameters (Pulse width, Repetition Rate (RR), Intensity). Static and dynamic targets, will appear on the screen at random locations and the subject will be instructed to response by aiming a narrow light beam at the targets on the screen. A CCD camera will capture the screen scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Systemically and visually Healthy (per history)
* Signed Informed Consent

Exclusion Criteria:

* Pregnant women
* Unwilling to sign informed consent
* Current and past history of migraine
* Current and post history of epilepsy or seizures
* Any known ocular disease in one or two eyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
visual cognition | instantaneous
  response time to targets after flashes

CONTACTS AND LOCATIONS:
Overall Officials: Shiri Soudry, DR, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Department of Ophthalmology, Rambam hospital, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided